CLINICAL TRIAL: NCT02606890
Title: Is the Lesion Pattern on Magnetic Resonance Imaging in Acute Ischemic Stroke Patients Associated With Atrial Fibrillation?
Brief Title: Stroke Lesion Pattern on MRI and Atrial Fibrillation
Acronym: SLPAF
Status: Completed | Type: Observational
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: Principal Investigator, Christian Nolte, Consultant, OA PD Dr. med., Charite University, Berlin, Germany
Other Study IDs: AGNO_001
Record Dates: First submitted 2015-11-13; First posted 2015-11-17 (Estimated); Last update posted 2016-12-08 (Estimated); Status verified 2016-12

CONDITIONS: Stroke; Atrial Fibrillation
Keywords: Magnetic Resonance Imaging; Stroke Lesion Pattern; Atrial Fibrillation; Stroke
MeSH Terms: conditions — Stroke; Atrial Fibrillation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: MRI — Stroke patients routinely undergo MRI at Charite Campus Benjamin Franklin. Type of MRI stroke pattern is evaluated with regard to presence or detection of (new) atrial fibrillation.

SUMMARY:
The aim of this retrospective cohort study is to investigate the relationship between lesion pattern on Magnetic Resonance Imaging (MRI) and atrial fibrillation in patients with acute ischemic stroke. The investigators hypothesize that a pattern with lesions located in at least two of the main arterial territories of the brain (left or right internal carotid artery or posterior circulation territory) is associated with atrial fibrillation.

The investigators will retrospectively analyze clinical data and imaging lesion pattern of 1000 consecutive patients who were admitted to the Department of Neurology (Charite - Universitätsmedizin Berlin, Campus Benjamin Franklin) and diagnosed with acute ischemic stroke.

Acute stroke patients of this cohort underwent 3-Tesla MRI with Diffusion-weighted Imaging (DWI) and Fluid-attenuated Inversion Recovery (FLAIR) sequences as well as standard 12-lead electrocardiography (ECG) on admission and cardiac monitoring with automated arrhythmia detection during stroke unit care lasting at least 24 hours.

If DWI and FLAIR lesions are located in more than one of the main arterial territories, lesion pattern will be categorized as "multiple lesion pattern".

The investigators hypothesize that a multiple lesion pattern will be detected more frequently in acute stroke patients with atrial fibrillation than in patients without atrial fibrillation.

The findings of this study might help to identify patients who could profit from extended diagnostic work-up in order to detect atrial fibrillation.

DETAILED DESCRIPTION:
Introduction

Atrial fibrillation is the most common cause of cardioembolic stroke and can be detected in about 27% of acute stroke patients treated on stroke units in Berlin. Stroke patients in whom atrial fibrillation is detected benefit from anticoagulation rather than anti-aggregation as a secondary prevention treatment. Lesions on brain imaging that are located in more than one of the main arterial territories of the brain may indicate cardioembolic etiology. Cardioembolic etiology is mainly due to atrial fibrillation. Atrial fibrillation causes cardiac emboli that may embolize in all brain arteries while other embolic sources e.g. carotid plaque cannot. However, current data on the association between lesion patterns and atrial fibrillation are inconclusive.

Purpose

The aim of this retrospective cohort study is to investigate the relationship between lesion pattern on Magnetic Resonance Imaging (MRI) and atrial fibrillation. The investigators hypothesize that a lesion pattern with brain lesions in more than one of the main arterial territories of the brain (left or right internal carotid artery or posterior circulation territory) is associated with atrial fibrillation in patients with acute ischemic stroke. The findings of this study might help to identify patients with atrial fibrillation.

Methods

Blinded for clinical data the investigators will analyze imaging data and radiologic reports of 1000 consecutive stroke patients who received 3-Tesla MRI imaging including Diffusion-weighted Imaging (DWI) and Fluid-attenuated Inversion Recovery (FLAIR) sequence. DWI lesions correspond to acute stroke and FLAIR lesions to subacute and chronic stroke. Brain lesions will be attributed to a vascular territory (left or right internal carotid artery or posterior circulation territory) and the pattern consecutively categorized as "single", "scattered" and "multiple" as described by Braemswig et al..

Fetal origin of the posterior cerebral artery and variability of vascular territories will be taken into account. Vascular territory attribution in ambiguous cases will be conducted by consensus between investigators. Demographic and clinical data will be collected from medical records. Strokes meeting the criteria for Embolic Stroke of Unknown Source (ESUS) will be identified according to Hart et al..

Based on a pilot study including 250 patients the investigators estimate that atrial fibrillation will be present in 38% of patients with a multiple lesion pattern on MRI and in 28% of patients with a non-multiple pattern. Based on these assumptions, 894 patients are required to have a 80% chance of detecting, (as significant at the 5% level), a difference of 10% with 28% atrial fibrillation in patients without multiple lesion pattern and 38% atrial fibrillation in patients with a multiple lesion pattern.

In accordance with legislation in Berlin, Germany, an ethics committee approval is not required for this study.

Outcomes

Primary outcome is multiple lesion pattern on MRI (DWI and FLAIR). Secondary Outcome is multiple lesion pattern on MRI (DWI lesions only) Analyses will be conducted comparing

* Patients with and without atrial fibrillation
* Patients with newly diagnosed atrial fibrillation and patients without atrial fibrillation
* Patients with newly diagnosed atrial fibrillation and patients with known atrial fibrillation
* Patients fulfilling ESUS criteria and patients who do not
* Patients with brain lesions outside of the overlap area of the main vascular territories as defined by Tatu et al.

ELIGIBILITY:
Inclusion Criteria:

* Acute ischemic stroke, defined as the presence of at least one DWI lesion and clinical signs of stroke
* underwent cerebral MRI imaging: DWI (diffusion-weighed imaging), FLAIR (Fluid-attenuated Inversion Recovery)
* admission to stroke unit at the Department of Neurology, Charite Campus Benjamin Franklin

Exclusion Criteria:

* unable to undergo MRI
* lack of data on heart rhythm

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with acute ischemic stroke proven by MRI admitted to Department of Neurology, Charite Campus Benjamin Franklin
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Actual)
Dates: Start 2015-08; Primary Completion 2016-10 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Lesion pattern on Magnetic Resonance Imaging in acute stroke patients | within 7 days after stroke onset
  Stroke lesion pattern on MRI is assessed.

SECONDARY OUTCOMES:
Lesion pattern on Magnetic Resonance Imaging in acute stroke patients (DWI only) | within 7 days after stroke onset
  Stroke lesion pattern on MRI is assessed (DWI only)

CONTACTS AND LOCATIONS:
Overall Officials: Christian H Nolte, PD Dr. med., Principal Investigator — Center for stroke Research Berlin, Charite-Universitätsmedizin, Berlin, Germany

REFERENCES:
- [Background] Bernstein RA, Di Lazzaro V, Rymer MM, Passman RS, Brachmann J, Morillo CA, Sanna T, Thijs V, Rogers T, Liu S, Ziegler PD, Diener HC. Infarct Topography and Detection of Atrial Fibrillation in Cryptogenic Stroke: Results from CRYSTAL AF. Cerebrovasc Dis. 2015;40(1-2):91-6. doi: 10.1159/000437018. Epub 2015 Jul 11. PMID 26182860
- [Background] Braemswig TB, Usnich T, Albach FN, Brunecker P, Grittner U, Scheitz JF, Fiebach JB, Nolte CH. Early new diffusion-weighted imaging lesions appear more often in stroke patients with a multiple territory lesion pattern. Stroke. 2013 Aug;44(8):2200-4. doi: 10.1161/STROKEAHA.111.000810. Epub 2013 Jun 13. PMID 23765944
- [Background] Hart RG, Diener HC, Coutts SB, Easton JD, Granger CB, O'Donnell MJ, Sacco RL, Connolly SJ; Cryptogenic Stroke/ESUS International Working Group. Embolic strokes of undetermined source: the case for a new clinical construct. Lancet Neurol. 2014 Apr;13(4):429-38. doi: 10.1016/S1474-4422(13)70310-7. PMID 24646875
- [Background] Kang DW, Chalela JA, Ezzeddine MA, Warach S. Association of ischemic lesion patterns on early diffusion-weighted imaging with TOAST stroke subtypes. Arch Neurol. 2003 Dec;60(12):1730-4. doi: 10.1001/archneur.60.12.1730. PMID 14676047
- [Background] Koennecke HC, Belz W, Berfelde D, Endres M, Fitzek S, Hamilton F, Kreitsch P, Mackert BM, Nabavi DG, Nolte CH, Pohls W, Schmehl I, Schmitz B, von Brevern M, Walter G, Heuschmann PU; Berlin Stroke Register Investigators. Factors influencing in-hospital mortality and morbidity in patients treated on a stroke unit. Neurology. 2011 Sep 6;77(10):965-72. doi: 10.1212/WNL.0b013e31822dc795. Epub 2011 Aug 24. PMID 21865573
- [Background] Saxena R, Koudstaal PJ. Anticoagulants for preventing stroke in patients with nonrheumatic atrial fibrillation and a history of stroke or transient ischaemic attack. Cochrane Database Syst Rev. 2004;2004(2):CD000185. doi: 10.1002/14651858.CD000185.pub2. PMID 15106146
- [Background] Tatu L, Moulin T, Vuillier F, Bogousslavsky J. Arterial territories of the human brain. Front Neurol Neurosci. 2012;30:99-110. doi: 10.1159/000333602. Epub 2012 Feb 14. PMID 22377874